CLINICAL TRIAL: NCT04306471
Title: Effect of Evolocumab in Patients With Critical Limb Ischemia
Brief Title: Effect of Evolocumab in Patients With Critical Limb Ischemia (Evol-CLI)
Acronym: Evol-CLI
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Leonardo Clavijo (Other)
Collaborators: Amgen (Industry)
Responsible Party: Sponsor-Investigator, Leonardo Clavijo, Associated Professor Cardiology, USC. Director Vascular Medicine and Peripheral Interventions Program Director, Interventional Cardiology Fellowship, University of Southern California
Organization: University of Southern California (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 20187090; HS-18-01010 (Other: Institutional Review Board)
Record Dates: First submitted 2020-02-21; First posted 2020-03-13 (Actual); Last update posted 2020-03-13 (Actual); Status verified 2020-03

CONDITIONS: Critical Limb Ischemia
Keywords: CLI, Gangrene, Ischemia, Amputation
MeSH Terms: conditions — Chronic Limb-Threatening Ischemia; Gangrene; Ischemia | interventions — evolocumab

STUDY DESIGN:
Intervention Model Description: This is a double-blinded, prospective, randomized, pilot, study
Who Masked: Participant, Care Provider, Investigator
Masking Description: Study subjects will be randomized, to receive either evolocumab or placebo. Each participant will have equal chance of receiving evolocumab or placebo. The study participant, the care provider and the investigator will not know to which study arm the participant was assigned.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Treatment arm (Experimental): 16 Patients with Critical Limb Ischemia on maximum statin therapy will receive in addition the study intervention involving a monthly subcutaneous injection of evolocumab 420 mg for 12 months
  Interventions: Drug: Evolocumab 140mg/mL Injector 1milliliter (mL) Pen x 3 for a monthly dose of 420 mg for 12 months.
- Control arm (Placebo Comparator): 16 Patients with Critical Limb Ischemia on maximum statin therapy will receive in addition a Placebo subcutaneous injection for 12 months.
  Interventions: Other: Placebo 1 milliliter (mL) Injector Pen x 3 monthly for 12 months

INTERVENTIONS:
Drug: Evolocumab 140mg/mL Injector 1milliliter (mL) Pen x 3 for a monthly dose of 420 mg for 12 months. — The study subjects randomized to the treatment study arm will receive monthly subcutaneous injections of evolocumab 420 mg in the abdomen, thigh or upper arm. The study drug (evolocumab) prefilled injector pens are to be provided by Amgen.
  Other Names: Repatha
  Arms: Treatment arm
Other: Placebo 1 milliliter (mL) Injector Pen x 3 monthly for 12 months — The study subjects randomized to the control study arm will receive monthly subcutaneous injections of placebo 1 mL x 3 in the abdomen, thigh or upper arm. The study placebo prefilled injector pens are to be provided by Amgen.
  Other Names: Control
  Arms: Control arm

SUMMARY:
Critical limb ischemia (CLI), is the most severe form of peripheral arterial disease (PAD), and clinically is characterized by pain at rest or non-healing ulcers of the lower extremities. Also, is associated with increased risk of cardiovascular death, myocardial infarction (MI), stroke and amputation.

Feringa et al. demonstrated in a study of 1,374 patients with PAD that all cause and cardiac related mortality rates were lower in patients at higher statin dose and lower levels of low-density lipoprotein cholesterol (LDL).

Patients with CLI statin therapy and lower LDL levels improve amputation-free survival and patency after revascularization procedures.

In the FOURIER trial, LDL cholesterol reduction with the PCSK9 inhibitor evolocumab in patients with symptomatic PAD with or without prior myocardial infarction or stroke was associated with improved major adverse cardiac events (MACE) and major adverse limb events (MALE) at 2-years.

The effect of evolocumab in patients with CLI , after a recent arterial revascularization and active wounds is not known, also it is not known whether the cholesterol lowering effect of evolocumab in this group of patients is equivalent to that of non-CLI PAD patients and what the effect is on arterial perfusion, wound healing and other biological markers of vascular physiology.

This study aims to investigate the effect of evolocumab in patients with CLI on maximally tolerated lipid lowering therapy with a statin for one year after an index CLI event, requiring revascularization.

DETAILED DESCRIPTION:
This is a double-blinded, prospective, randomized, pilot, study in thirty-two subjects with clinical CLI on background treatment with a statin. Subjects will be assessed based on their medical history and physical examination. Eligible subjects must meet all inclusion criteria and none of the exclusion criteria. There will be a treatment group and a placebo group, each with equal number of participants (n=16 patients in each group). After consent and enrollment, subjects will have a venous blood sample drawn to perform a lipid profile, serum vascular growth factors such as: vascular endothelial growth factor (VEGF), soluble VEGF receptor-1 (sVEGFR-1), soluble VEGF receptor-2 (sVEGFR-2), fibroblast growth factor (FGF), von Willebrand factor (vWF), tissue plasminogen activator (TPA) and plasminogen activator inhibitor -1 (PAI-1) and endothelial progenitor cells (EPCs). The investigators will then perform lower extremity arterial perfusion assessment of the affected and unaffected limb as rest ankle-brachial index (ABI), toe-brachial index (TBI), bilateral transcutaneous partial pressure of oxygen (TcPO2), spatial frequency domain imaging (SFDI), femoral studies (FMT, compliance, distensibility and stiffness), brachial endothelial function testing (FMD after hyperemia and maximal vasodilation). The study participant subjects will receive monthly subcutaneous injections of evolocumab 420 mg or placebo injections.

The LDL cholesterol will be measured at the baseline and a blinded measurement will also be performed at 3 and 12 months.

In patients with active wounds, healing will be evaluated at baseline and every month for six months by photographic analysis using planimetry and 2D/3D topographic analysis.

The study participants patients will be seen at 3, 6, and 9 months for follow up.

After 12 months +/- 2 weeks, all tests will be repeated.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent.
* Age ≥40 to ≤85 years of age at the time of consent.
* Diagnosis CLI, Rutherford class IV to VI at the time of diagnosis, toe pressure ≤30 mmHg in non-diabetics or ≤40 mmHg in diabetics, angiography, duplex ultrasound or history of lower extremity surgical or endovascular revascularization for CLI.
* Stable on maximal tolerated dose of a statin, defined as the highest dose of statin (preferably atorvastatin or rosuvastatin) tolerated by the patient without side effects for at least one month.

Exclusion Criteria:

* Less than 1 month from last revascularization procedure including surgery or endovascular procedures.
* Subjects with active infection.
* Diabetes therapy with canagliflozin
* Subjects who in the opinion of the Principal Investigator will likely require additional. amputation or revascularization procedures during the duration of the study.
* Subjects with anticipated need of cardiac or surgical revascularization procedures.
* Subjects with chronic inflammatory conditions or requiring chronic systemic corticosteroids.
* New York Heart Association (NYHA) class III or IV heart failure, or known left ventricular ejection fraction <30%.
* Uncontrolled arrhythmia.
* Uncontrolled hypertension with systolic BP>180 mmHg or diastolic >100 mmHg.
* Untreated thyroid disease.
* Severe chronic renal disease with estimated glomerular filtration rate (eGFR) <20 mL/min.
* Liver disease with aspartate aminotransferase (AST) or alanine aminotransferase (ALT) ≥3 times the upper limit of normal.
* Status post-organ transplant.
* Pregnant and breastfeeding women.
* Fertile age female not on appropriate birth control.
* Clinically significant disease that, in the opinion of the Principal Investigator, is likely to require surgery or immunotherapy that may interfere with the completion of the study.
* Active cancer or life expectancy of less than two years.
* Chronic anticoagulation or hypercoagulability disorder.
* Atrial fibrillation with a CHADS-VASc Score ≥2 or any clinical condition which, in the opinion of the Principal Investigator increases the risk of cerebrovascular events.

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2020-02-24 (Actual); Primary Completion 2021-02-04 (Estimated); Study Completion 2022-02-04 (Estimated)

PRIMARY OUTCOMES:
Evolocumab effect on LDL cholesterol changes in patients with Critical Limb Ischemia | 3 months
  To evaluate LDL cholesterol values in mg/dL in patients with Critical Limb Ischemia at baseline and after receiving three month therapy of Evolocumab compared to placebo.
  The LDL cholesterol value changes will be measured as least-squares mean percentage

SECONDARY OUTCOMES:
Evolocumab effect on Lower extremity arterial perfusion changes on ankle-brachial indices (ABI). | 12 months
  To evaluate lower extremity arterial perfusion of the affected and unaffected limb in patients with CLI at baseline and after a 12 month therapy with evolocumab, measured by rate changes in ankle-brachial indices (ABI).
  The ABI will be determined by the dorsalis pedis and posterior tibialis arteries highest systolic pressure value (in mmHg) of each foot divided by the brachial artery highest systolic pressure (in mmHg) of both arms.
Evolocumab effect on Lower extremity arterial perfusion pressure changes on toe-brachial indices (TBI). | 12 months
  To evaluate lower extremity arterial perfusion of the affected and unaffected limb in patients with CLI at baseline and after a 12 month therapy with evolocumab, measured by rate changes in toe-brachial indices (TBI).
  The TBI will be determined by the great toe pressure (in mmHg) of each foot divided by the brachial artery highest systolic pressure (in mmHg) of both arms.
Evolocumab effect on Lower extremity microvascular perfusion changes. | 12 months
  To evaluate lower extremity microvascular perfusion of the affected and unaffected limb in patients with CLI at baseline and after a 12 month therapy with evolocumab compared with placebo, measured by tcpo2 mmHg changes in transcutaneous oxygen tension in the skin.
  Transcutaneous oxygen will be performed by placing electrodes on the skin at different levels of each leg, foot and chest for reference.
Evolocumab effect on foot perfusion changes. | 6 months
  To evaluate transcutaneous oxy-hemoglobin and deoxy-hemoglobin foot perfusion of the affected and unaffected foot in patients with CLI at baseline and after 6 month therapy with evolocumab compared with placebo, assessed by spatial frequency domain imaging (SFDI) mapping changes measured in percentage %.
  Transcutaneous oxy-hemoglobin and deoxy-hemoglobin will be performed by obtaining SFDI images on the skin at different levels of each foot.
Evolocumab effect on Femoral arterial distensibility changes. | 12 months
  To evaluate common femoral artery distensibility of the affected and unaffected limb in patients with CLI at baseline and after 12 month therapy with evolocumab compared with placebo, measured by the relative change in lumen area during systole for a given pressure change ( 10-3 x kPa-1).
  Femoral distensibility will be performed by correlating systemic blood pressure and continuously recording by linear ultrasound using a LOGIQ eR7 ultrasound and a 12-L-RS linear array transducer and images analyzed by the QUIPU automated cardiovascular suite, carotid studio imaging software.
Evolocumab effect on Femoral artery Medial Thickness (FMT) changes. | 12 months
  To evaluate common femoral artery medial thickness changes of the affected and unaffected limb in patients with CLI at baseline and after 12 month therapy with evolocumab compared with placebo.
  The common femoral artery medial thickness will be measured in millimeters (mm) and performed by correlating systemic blood pressure and continuously recording by linear ultrasound using a LOGIQ eR7 ultrasound and a 12-L-RS linear array transducer and images analyzed by the QUIPU automated cardiovascular suite, carotid studio imaging software.
Evolocumab effect on endothelial function by Flow Mediated Dilation (FMD) changes. | 12 months
  To evaluate brachial artery flow mediated dilation (brachial artery diameter in response to shear stress) of both arms in patients with CLI, at baseline and after 12 month therapy with evolocumab compared with placebo.
  The FMD will be measured as the percentage (%) change in brachial artery diameter from baseline in response to the increase flow achieved after the inflation of a pneumatic cuff to supra-systolic pressure for 5 minutes The ultrasound brachial images will be acquired using a LOGIQ eR7 ultrasound and a 12-L-RS linear array transducer. Images will be analyzed by the QUIPU automated cardiovascular suite, FMD studio imaging software.

OTHER OUTCOMES:
Evolocumab effect on wound healing changes. | 6 months
  To evaluate wound healing of the affected lower limb in patients with CLI at baseline and after 6 month therapy with evolocumab compared with placebo, assessed by wound size planimetry and wound 2D/3D topographic analysis in millimeters (mm).
Evolocumab effect on serum levels of vascular endothelial growth factors changes. | 12 months
  To evaluate serum levels of vascular endothelial growth factor receptors 1 and 2 (sVEGFR-1 and sVEGFR-2) in patients with CLI at baseline and after 12 month therapy with evolocumab compared with placebo, measured in pg/ml using quantitative sandwich ELISA.
Evolocumab effect on circulating endothelial progenitor cells changes | 12 months
  To evaluate circulating endothelial progenitor cells (EPCs) in patients with CLI at baseline and after 12 month therapy with evolocumab compared with placebo.
  The number of EPCs will be determined by flow cytometry (FACs) analysis. For fluorescent activated cell-sorting analysis, mononuclear cells will be resuspended in phosphate buffer saline (PBS), 0.1% bovine albumin and aprotinin (20µ/mL). Immunofluorescent staining will be performed by incubating with fluorescent conjugated antibody CD-34 fluorescein isothiocyanate (FITC), kinase insert domain receptor (KDR) and CD133-phycoerythrin (PE).
  Cell fluorescence will be measured immediately after staining.

CONTACTS AND LOCATIONS:
Overall Officials: Leonardo Clavijo, MD, PhD, Principal Investigator — University of Southern California
Locations (1):
- University of Southern California, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No